CLINICAL TRIAL: NCT06744946
Title: Comparison Between Pleurodesis by a Combination of Bleomycin and Tranxemic Acid Solution and Thoracoscopic Talc Poudrage in Malignant Pleural Effusion
Brief Title: Thoracoscopic Talc Pleurodesis Versus Bleomycin -Tranxemic Acid Mixture Injection in Chest Tube in Malignant Pleural Effusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mohamed Sabry (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Mohamed Sabry, Lecturer of chest diseases, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Talc Pleurodesis - Bleomycin
Record Dates: First submitted 2024-12-07; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Malignant Pleural Effusions (Mpe)- Pleurodesis; Pleurodesis
Keywords: Talc -pleurodesis-bleomycin
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — Thoracoscopes

STUDY DESIGN:
Intervention Model Description: comparing between two groups of thirty patients each,the first group will include talc poudrage pleurodesis and the second include chest tube injection of a mixture of bleomycin and tranxemic acid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- the first arm thoracoscopic talc poudrage and the second arm Bleomycin -Tranxemic mic acid mixture (Experimental): the first arm is talc insufflation through medical thoracoscopy the second arm involve bleomycin- tranxemic acid mixture injection in intercostal tube
  Interventions: Procedure: thoracoscope

INTERVENTIONS:
Procedure: thoracoscope — bleomycin- tranxemic acid mixture pleurodesis versus thoracoscopic talc poudrage
  Other Names: intercostal tube

SUMMARY:
Comparing Two Methods to Treat Fluid Build-up in Chest for Cancer Patients:Talc Powder Surgery versus Chest Tube Medicine.

DETAILED DESCRIPTION:
Closure of the space where the effusion is recurrently accumulated through talc poudrage in thoracoscopy or bleomycin - tranxemic acid solution injection in chest tube.

ELIGIBILITY:
Inclusion Criteria:

- 1. Adult patients (more than 18 years) with malignant pleural effusion or highly suspected exudate.

2. Fit patients for the procedure selected.

Exclusion Criteria:

1. Inability to provide informed consent for the procedure.
2. Hemodynamically unstable patients.
3. Bleeding diathesis.
4. Uncontrolled cough.
5. Hypoxic index less than 300.
6. Endobronchial obstruction.
7. Pleural thickening with trapped lung.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Dyspnea Borg Scale | one month
  the rate of shortness of breath from number 0 to number 10

CONTACTS AND LOCATIONS:
Overall Officials: mohamed sabry eltarhony, lecturer, Principal Investigator — Alexandria University
Locations (1):
- Chest Department -Faculty of Medicine, Alexandria, Azarita, Egypt

IPD SHARING:
Plan to Share IPD: No
because the facility, where i do my work, refuse to share any project untill it is fully published

REFERENCES:
- See also: Safety of pleurodesis with talc poudrage in malignant pleural effusion: a prospective cohort study. Lancet . 2007 May 5;369(9572):1535-1539 — https://pubmed.ncbi.nlm.nih.gov/17482984/
- Available data/document: Study Protocol: msabry776@yahoo.com — https://pubmed.ncbi.nlm.nih.gov/17482984/ — very good